CLINICAL TRIAL: NCT05660733
Title: French Registry Studying the Characteristics and Prognosis of Aortic and Large Arterial Vessel Infections
Brief Title: Study of the Aortic and Large Arterial Vessel Infections
Acronym: Repia
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: Research on existing data
Record Dates: First submitted 2022-12-07; First posted 2022-12-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Aortic Infections and Inflammations; Mycotic Aneurysm; Arterial Infections and Inflammations; Prosthetic Infection
MeSH Terms: conditions — Inflammation; Aneurysm, Infected

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aortic or large arterial vessel infections are rare but serious infections. Their management is based on French and American expert opinions. The quality of evidence supporting these guidelines is low because most publications on the subject correspond to case series and few interventional studies have been performed to validate their management. However, referral centres for vascular surgery are frequently solicited to give their opinion on patients suffering from mycotic aneurysms. In addition, the last few decades have seen the improvement of vascular surgery techniques allowing the management of more and more patients, often elderly and comorbid. There has therefore been an increase in the incidence of infectious complications associated with this care. It is therefore essential to participate in research on aortic and large arterial vessel infections. For this, a monocentric cohort study seems to be an essential first step to better understand the polymorphism and complexity of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Aortic or large arterial vessel infection. The diagnosis is made on a number of criteria in favour of the diagnosis (at least 2 of the following 3 criteria):

  * Compatible clinical presentation: local or general inflammatory signs suggestive of a deep infection (fever, chills, scar discharge, fistula, febrile abdominal pain and low back pain, ...) or per-operative finding of an infection in contact with native or prosthetic vascular tissue
  * And/or biological (inflammatory syndrome) and/or imaging evidence (infectious sign on native, bioprosthetic or prosthetic vascular tissue on CT and/or PET scan) in favour of the diagnosis
  * And/or microbiological evidence (positive serologies, blood cultures or deep samples in favour of infection)

Exclusion Criteria:

* Patient who objected to participation in this protocol and data collection
* Pregnant woman, parturient or breastfeeding mother
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care by virtue of articles L.3212-1 and L.3213-1 of the French public health code
* Person subject to a legal protection measure
* Person unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patients with proved aortic or large arterial vessel infection and without exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
one-year mortality | one year after the diagnosis
  Study of all-cause mortality in patients with aortic vascular infection and large arterial vessels during the first year of follow-up after diagnosis.

SECONDARY OUTCOMES:
Identification of prognostic factors associated with arterial vascular infections | at the time of diagnosis and up to one year afterwards
  Identification of prognostic factors in patients with aortic and large arterial vessel infection: a multivariate Cox model to identify factors associated with mortality or better survival

CONTACTS AND LOCATIONS:
Overall Officials: Lefèvre Benjamin, M.D., Principal Investigator — Université de Lorraine & CHRU de Nancy
Locations (1):
- Université de Lorraine, CHRU Nancy and APEMAC, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lalevee L, Serguei M, Jeanbert E, Simon M, Luc A, Settembre N, Henard S, Novy E, Guerci P, Lefevre B. Characteristics and outcomes of patients with infective native aortic aneurysm or vascular graft and endograft infection. Infect Dis (Lond). 2025 Oct;57(10):920-932. doi: 10.1080/23744235.2025.2502826. Epub 2025 May 16. PMID 40377031